CLINICAL TRIAL: NCT00574145
Title: Examining the Effect of Healing Touch on Radiotherapy-induced Fatigue
Brief Title: Healing Touch in Treating Fatigue in Women Undergoing Radiation Therapy for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nancy Wells, Research Professor of Nursing; Director, VUMC Nursing, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC SUPP 0633; VU-VICC-SUPP-0633
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer; Depression; Fatigue
Keywords: fatigue; depression; psychosocial effects of cancer and its treatment; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Depression; Fatigue | interventions — Therapeutics; Psychiatric Rehabilitation; Therapeutic Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy/Supportive Care (A) (Experimental): Patients receive radiotherapy and healing touch therapy from a healing touch therapist once a week for the duration of their radiotherapy
  Interventions: Procedure: Bio-field energy therapy; Procedure: fatigue assessment and management; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment; Procedure: therapeutic touch
- Control ARM (B) (Sham Comparator): Patients receive radiotherapy and sham healing touch therapy from a sham healing touch therapist once a week for the duration of their therapy
  Interventions: Procedure: fatigue assessment and management; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: Bio-field energy therapy — Practitioner's hands to influence the human energy field surrounding the patient's body.
  Other Names: biofield therapy
  Arms: Radiotherapy/Supportive Care (A)
Procedure: fatigue assessment and management — duration
Procedure: psychosocial assessment and care — duration
Procedure: quality-of-life assessment — duration
Procedure: therapeutic touch — Practitioner's hands to influence the human energy field surrounding the patient's body
  Arms: Radiotherapy/Supportive Care (A)

SUMMARY:
RATIONALE: Healing touch therapy may be effective in lessening fatigue in women with breast cancer who are undergoing radiation therapy.

PURPOSE: This randomized clinical trial is studying how well healing touch works in treating fatigue in women undergoing radiation therapy for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the ability to recruit and retain patients with breast cancer receiving curative radiotherapy in a Complementary and Alternative Medicine trial.
* To determine the acceptability of weekly healing touch therapy to patients with breast cancer who receive curative radiotherapy.
* To examine the effect of healing touch on fatigue and quality of life for patients with breast cancer receiving radiotherapy as a component of therapy.

OUTLINE: Patients are stratified by type of treatment (radiotherapy alone vs chemotherapy completed prior to radiotherapy)

* Arm I:Patients receive healing-touch therapy administered once a week for 45 minutes by a healing-touch therapist for the duration of radiotherapy.
* Arm II: Patients receive sham-therapy administered once a week for 45 minutes by a sham-practitioner (NOT a healing-touch therapist) for the duration of radiotherapy.

Patients complete the Hospital Anxiety and Depression Scale (HAD) and a demographic variables form (age, race/ethnicity, marital status, employment) at baseline. Patient fatigue is measured on a weekly basis throughout radiotherapy with completion of the Brief Fatigue Inventory (BFI). The Functional Assessment of Cancer Therapy-Breast form (FACT-B) is completed at baseline and the end of radiotherapy. Patients undergo a 20-minute interview at the end of study to determine the acceptability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven breast cancer
* Receiving post lumpectomy or post mastectomy radiation therapy (RT)
* Eastern Cooperative Oncology Group performance status of 0, 1 or 2
* Prescribed a minimum of 5 weeks of RT
* Between the ages of 21 and 75
* Able to speak English.
* Provides written informed consent

Exclusion Criteria:

* Documented active psychiatric illness
* Documented cognitive impairment that would preclude the ability to provide informed consent.
* Stage IV breast cancer
* Receiving concurrent chemotherapy and RT

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Wells, DNSc, RN, Principal Investigator — Vanderbilt-Ingram Cancer Center; Fern Fitzhenry, PhD, RN, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] FitzHenry F, Wells N, Slater V, Dietrich MS, Wisawatapnimit P, Chakravarthy AB. A randomized placebo-controlled pilot study of the impact of healing touch on fatigue in breast cancer patients undergoing radiation therapy. Integr Cancer Ther. 2014 Mar;13(2):105-13. doi: 10.1177/1534735413503545. Epub 2013 Oct 7. PMID 24105358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled February 2007 to March 2009.
Pre-assignment Details: Forty-four patients signed consent, all were eligible.
Groups:
- Control ARM (B): Patients receive radiotherapy and sham healing touch therapy from a sham healing touch therapist once a week for the duration of their radiotherapy
Period: Overall Study
Arm/Group | Radiotherapy/Supportive Care (A) | Control ARM (B)
Started | 22 | 22
Completed | 20 | 21
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiotherapy/Supportive Care (A) | Control ARM (B) | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 50 (1) | 51 (1) | 51 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Using the Brief Fatigue Inventory (BFI)
Description: 9-items with an 11-point rating scale measures intensity of fatigue (3 items, 0 = no fatigue to 10 = fatigue as bad as you can imagine) and interference of fatigue on daily life (6 items, 0 = does not interfere to 10 = completely interferes. Each participant's score is summed with a possible minimum score of 0 and a possible maximum score of 90. A mean score was then determined.
Time Frame: 6 weeks
Population: Patients who completed 5 of 8 maximum collection points. Arm A: 1 patient withdrew at 2 days, 1 patient withdrew at 5 days. Arm B: 1 patient withdrew at 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Radiotherapy/Supportive Care (A): Patients receive radiotherapy and healing touch therapy from a healing-touch therapist once a week for the duration of their radiotherapy
- Control ARM (B): Patients receive radiotherapy and sham healing touch therapy from a sham healing-touch therapist once a week for the duration of their radiotherapy
Arm/Group | Radiotherapy/Supportive Care (A) | Control ARM (B)
Number analyzed (Participants) | 20 | 21
units on a scale | 2.786 (0.1963) | 1.356 (0.1413)

2. Secondary Outcome: Quality of Life as Measured by the Functional Assessment of Cancer Therapy-Breast Form (FACT-B)
Description: 36 items that measure general quality of life (27 items) and specific breast cancer concerns (9 items) on a 5-point rating scale with 0 = not at all to 4 = very much. Minimum (worst quality of life) possible score = 0 and maximum (best quality of life) possible score = 144. Physical and emotional well-being scores were reverse coded and sub scale scores were summed. Median scores for baseline and at 6 weeks were determined
Time Frame: baseline and 6 weeks
Population: Arm A:1 patient was accidentally notified of group assignment before final data collected, 2 patients withdrew (1 at 2 days), 1 at 5 days. )Arm B: 1 patient withdrew at 4 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Radiotherapy/Supportive Care (A) | Control ARM (B)
Number analyzed (Participants) | 20 | 21
units on a scale
  Baseline | 61 [50 to 85] | 65 [54 to 76]
  6 Weeks | 65 [44 to 76] | 67 [44 to 77]

3. Secondary Outcome: Intensity of Anxiety and Depression
Description: Measured on the Hospital Anxiety and Depression Scale, 14 items on a 4-point scale scored from 0 = not at all (best feeling) to 3 = very often (worst feeling). Scores are summed and range from a minimum of 0 (no anxiety or depression) to 42 (worst anxiety or depression)and a median for each arm is determined at the specified timepoints.
Time Frame: baseline and off-radiation at 5 to 7 weeks
Population: Arm A: 1 patient withdrew at 2 days, 1 patient withdrew at 5 days. Arm B: 1 patient withdrew at 4 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Radiotherapy/Supportive Care (A) | Control ARM (B)
Number analyzed (Participants) | 20 | 21
units on a scale
  Baseline | 21 [16 to 28] | 23 [16 to 29]
  At 5 to 7 weeks | 28 [21 to 40] | 28 [21 to 37]

ADVERSE EVENTS:
Arm/Group | Radiotherapy/Supportive Care (A) | Control ARM (B)
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes